CLINICAL TRIAL: NCT05976477
Title: Reduction Of Dietary Salt Intake To Control Systolic Blood Pressure In Hypertensive Older Patients: The Repress Randomized Controlled Trial
Brief Title: Reduction Of Dietary Salt Intake To Control Systolic Blood Pressure In Hypertensive Older Patients
Acronym: REPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Principal Investigator, Carlotta Franchi, PRINCIPAL INVESTIGATOR, Mario Negri Institute for Pharmacological Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRFMN-REPRESS-ONFOODS
Record Dates: First submitted 2023-04-11; First posted 2023-08-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: randomized controlled trial; older patients; polypharmacy; diet; salt intake; educational intervention; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention arm during the 12 weeks after randomization will receive on their smartphone and/or via e-mail, information materials such as videos, images and recipes for reminders specifically designed to make patients aware on the importance of reducing dietary salt intake and suggestions on how to do it. The educational interventions will be delivered once a week. The main objective of the educational interventions is to spread knowledge about the health risks of excessive salt intake, the actual amount of salt in food, measures to reduce salt intake (e.g. use spices, eat fresh fruits and vegetables, check food labels, gradually reduce the salt in favorite recipes, avoid putting salt and salty sauces on the table, etc.). The interventions, conceived with nutritionists, will be delivered once a week to the participants and to their caregivers and/or the closest family member, involved in the food shopping and the preparation of meals.
  Interventions: Other: educational intervention
- Control (No Intervention): Patients randomized to Control Group will only receive short tips on controlling blood pressure.

INTERVENTIONS:
Other: educational intervention — 1. four short videos (about one-minute/one-minute and half duration) concerning the topic of reducing dietary salt intake to control the blood pressure in elderly hypertensive patients: the mini-videos will be designed with a common thread starting from providing general information regarding diet to enhance awareness of the amount of salt that is usually introduced with the diet, up to give suggestions on which products to choose/avoid during grocery shopping and how to behave during the preparation and consumption of food at home to reduce salt intake;
  2. Four images informing participants about the risk of excessive salt intake and health benefits of a low-sodium diet and tips on how to reduce daily salt intake;
  3. Four recipes for tasty easy-to-prepare meals, avoiding added salt.
  Arms: Intervention

SUMMARY:
REPRESS is an open label, pragmatic, multicenter, randomized controlled phase III trial with blinded endpoint with 1:1 (intervention to control arm) allocation ratio.

The REPRESS trial is aimed to determine the efficacy of an educational intervention aimed at reducing dietary salt intake in elderly people (60+) with moderate hypertension and exposed to polypharmacy (3+ drugs) in improving systolic BP control compared to an attention arm.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling patients aged ≥60 years;
2. Prescribed ≥3 drugs;
3. A) Systolic blood pressure ≥130 and ≤160 mmHg for patients prescribed stable antihypertensive therapy (at least 1 drug (ATC code: C02*, C03*, C07*, C08*, C09*)); B) Systolic blood pressure ≥140 and ≤160 mmHg for those patients not prescribed any antihypertensive drug;
4. Capable of feeding independently;
5. Own a smartphone;
6. Frequently consuming home-cooked meals (≥4 days during a week and ≥3 during the weekend per month);
7. Giving signed informed consent.

Exclusion Criteria:

1. Living in a nursing home or having applied for nursing home admission;
2. Being prescribed (adding, switching or changing dosage) an antihypertensive drug in the three months before enrollment;
3. Undergoing renal replacement therapy with dialysis or having renal impairment with estimated glomerular filtration rate (eGFR) <25 mL/min/1.73 m2 (assessed by CKD-EPI formula) [30] within previous six months or at the screening assessment;
4. Following a low-sodium dietary regimen;
5. Being unable or refusing to sign informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic BP | 6 months
  The primary outcome will be the change in systolic BP defined as the difference from baseline to 12 weeks follow-up in the two study groups.

SECONDARY OUTCOMES:
Change in 24-hour urinary sodium excretion | 6 and 12 months
  The change in the level of 24-hour urinary sodium excretion as the difference from baseline to 12 weeks follow-up (short follow-up), or 6 and 12 months (long follow-up) in the two study arms
Change in adherence to the mediterranean diet | 6 and 12 months
  The change in dietary habits of elderly patients during the 12 months follow-up in the two study groups measured by the adherence to Meditteranean Diet evaluated through the PREDIMED score (higher values correspond to better quality diet)
Incidence of cardio- and cerebro-vascular events | 12 months
  The difference in the incidence of cardio- and cerebro-vascular events during 12-months follow-up between the intervention and the control arm

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Franchi, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri